CLINICAL TRIAL: NCT04293666
Title: Functional Evaluation of Kefir Drink on Antifatigue and Improving Exercise Performance
Brief Title: Functional Evaluation of Kefir Drink on Antifatigue and Exercise Exercise Performance-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Sport University (Other)
Collaborators: Synbio Tech Inc. (Industry)
Responsible Party: Principal Investigator, Chi-Chang Huang, PI, National Taiwan Sport University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 00001
Record Dates: First submitted 2020-02-19; First posted 2020-03-03 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Exercise Performance; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Kefir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kefir drink (Experimental): (2) The first phase of Kefir, the second phase of the placebo group (hereinafter referred to as group B
  Interventions: Dietary Supplement: Kefir
- placebo (Placebo Comparator): (1) first-stage placebo and second-stage Kefir group (hereinafter referred to as group A).
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Kefir — 28 days supplementation kefir drink (prepared by inoculating pasteurized 9.2% reconstituted skim milk with powder kefir starter culture and fermented at 37 °C for 16 h. The fermented milk was then pasteurized at 100 °C for 30 min and freeze dried. The powder kefir starter culture used for inoculation was composed of defined lactic acid bacteria strains which contains Lactobacillus fermentum DSM 32784 (LF26), L. helveticus DSM 32787 (LH43), L. paracasei DSM 32785 (LPC12), L. rhamnosus DSM 32786 (LRH10), and Streptococcus thermophilus DSM 32788 (ST30)), 200ml/day
  Arms: Kefir drink
Dietary Supplement: placebo — Maltodextrin, same calorie as kefir, 200ml/day
  Arms: placebo

SUMMARY:
Purpose: The aim of the present study was to evaluate potential beneficial effects of Kefir drink (Synbio Tech Inc., Kaohsiung City, Taiwan) on fatigue and ergogenic functions following physiological challenge. Methods: 16 male subjects, 8 in each group, were divided into two groups according to the principle of maximal oxygen uptake, which were (1) first-stage placebo and second-stage Kefir group (hereinafter referred to as group A). (2) The first phase of Kefeier, the second phase of the placebo group (hereinafter referred to as group B), after 4 weeks of supplementation, the performance and fatigue resistance tests were carried out in sequence, including: treadmill aerobic endurance exhaustion time, and fixation Exercise time and intensity challenge changes in blood lactate, blood urea nitrogen concentration and creatine kinase activity, as well as differences in body composition before and after supplementation. After the first phase of the test is completed, the four weeks of emptying are performed. And after adding the crossover sample, perform four weeks of supplementation and testing again.

ELIGIBILITY:
Inclusion Criteria:

* >20 years old
* health

Exclusion Criteria:

* No smoking
* drinking habits
* no nutritional supplements or medications
* no food allergies
* normal liver and kidney function
* no diabetes and other chronic diseases

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-01-27 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Exercise endurance exhaustion time | 28 days
  We adopted a double-blind test in which the volunteers, based on their basal maximal oxygen consumption (VO2max). before and after intervention, the individual basal VO2max during pretest was used as a reference to adjust the individually appropriate exercise intensity to measure exhaustive endurance (85% VO2max) and recording the running time from begin to exhaust.
Clinical Biochemistry of lactate level | 28 days
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 5 (E5), 10 (E10), 15 (E15), and 30 (E30) min during the exercise phase, and 20 (R20), 40 (R40), 60 (R60), and 90 (R90) min in the recovery phase. Serum lactate (mmol/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Clinical Biochemistry of ammonia level | 28 days
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 5 (E5), 10 (E10), 15 (E15), and 30 (E30) min during the exercise phase, and 20 (R20), 40 (R40), 60 (R60), and 90 (R90) min in the recovery phase. Serum ammonia (umol/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Clinical Biochemistry of CK level | 28 days
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 5 (E5), 10 (E10), 15 (E15), and 30 (E30) min during the exercise phase, and 20 (R20), 40 (R40), 60 (R60), and 90 (R90) min in the recovery phase. Serum CK (U/L), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).
Clinical Biochemistry of glucose level | 28 days
  For assessment of fatigue-related indices, volunteers fasted for at least 8 h before the 60% VO2max fixed intensity exercise challenge. Blood samples were collected with an arm venous catheter at indicated time points during exercise and recovery periods, including baseline (0), 5 (E5), 10 (E10), 15 (E15), and 30 (E30) min during the exercise phase, and 20 (R20), 40 (R40), 60 (R60), and 90 (R90) min in the recovery phase. Serum glucose (mg/dL), were assessed for monitoring physiological adaptation. All biochemical indices were assessed using an autoanalyzer (Hitachi 7060, Tokyo, Japan).

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Sport University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No